CLINICAL TRIAL: NCT02682433
Title: 3D Sonohysterography vs Hysteroscopy: Study for the Evaluation of Intrauterine Abnormalities
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 522-15
Record Dates: First submitted 2016-01-12; First posted 2016-02-15 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Uterine Diseases
MeSH Terms: conditions — Uterine Diseases | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diagnostic hysteroscopy (Experimental): Women who were routinely referred to perform diagnostic hysteroscopy. As part of the procedure, clear liquid is inserted into the uterine cavity. After the hysteroscopy, and in the same position, abdominal and vaginal sonar will be performed, and the findings will be recorded and will be compared. Immediately after completion of the office hysteroscopy, two-dimensional and three-dimensional sonar to demonstrate the uterine cavity and its walls will be performed while using the liquid which is left in the uterine cavity. It is important to note that no additional invasive operation will be performed beyond what is necessary to perform hysteroscopy. It should be emphasized that the sonar test will be performed immediately and in the same position as the hysteroscopy test. All procedures will be performed in women clinics or day hospitalization. It should be noted that the medical examinations will not be performed unless there are medical reasons.
  Interventions: Device: diagnostic hysteroscopy
- diagnostic sonar test (Experimental): Women who were routinely referred to perform diagnostic hysteroscopy. As part of the procedure, clear liquid is inserted into the uterine cavity. After the hysteroscopy, and in the same positionabdominal and vaginal sonar will be performed, and the findings will be recorded and will be compared. Immediately after completion of the office hysteroscopy, two-dimensional and three-dimensional sonar to demonstrate the uterine cavity and its walls will be performed while using the liquid which is left in the uterine cavity. It is important to note that no additional invasive operation will be performed beyond what is necessary to perform hysteroscopy. It should be emphasized that the sonar test will be performed immediately and in the same position as the hysteroscopy test. All procedures will be performed in women clinics or day hospitalization. It should be noted that the medical examinations will not be performed unless there are medical reasons.
  Interventions: Device: diagnostic sonar test

INTERVENTIONS:
Device: diagnostic hysteroscopy — Women who were routinely referred to perform diagnostic hysteroscopy. As part of the procedure, clear liquid is inserted into the uterine cavity. After the hysteroscopy, abdominal and vaginal sonar will be performed, and the findings will be recorded and will be compared. Immediately after completion of the office hysteroscopy, two-dimensional and three-dimensional sonar to demonstrate the uterine cavity and its walls will be performed while using the liquid which is left in the uterine cavity. It is important to note that no additional invasive operation will be performed beyond what is necessary to perform hysteroscopy. It should be emphasized that the sonar test will be performed immediately and in the same position as the hysteroscopy test. All procedures will be performed in women clinics or day hospitalization. It should be noted that the medical examinations will not be performed unless there are medical reasons.
  Arms: diagnostic hysteroscopy
Device: diagnostic sonar test — Women who were routinely referred to perform diagnostic hysteroscopy. As part of the procedure, clear liquid is inserted into the uterine cavity. After the hysteroscopy, abdominal and vaginal sonar will be performed, and the findings will be recorded and will be compared. Immediately after completion of the office hysteroscopy, two-dimensional and three-dimensional sonar to demonstrate the uterine cavity and its walls will be performed while using the liquid which is left in the uterine cavity. It is important to note that no additional invasive operation will be performed beyond what is necessary to perform hysteroscopy. It should be emphasized that the sonar test will be performed immediately and in the same position as the hysteroscopy test. All procedures will be performed in women clinics or day hospitalization. It should be noted that the medical examinations will not be performed unless there are medical reasons.
  Arms: diagnostic sonar test

SUMMARY:
Uterine cavity diseases can cause mild to severe symptoms, and may indicate the functional problems of the female reproductive system. Many articles examine the efficacy of diagnostic hysteroscopy compared to sonohysterography in the diagnosis of uterine cavity diseases. Most of the articles are from the last decade, but the subject has been laid aside in the recent years. Antonio Simone Lagana and his group have found that there is 100% correlation in uterine cavity structure between diagnostic hysteroscopy and sonohysterography, and only 78% correlation when it comes to intrauterine fibroids and polyps. Walid El-Sherbiny, MD and his group have found that there is a significant advantage to three-dimensional sonohysterography over two-dimensional in the diagnosis of uterine cavity diseases. No significant difference was observed, and 97% correlation was found, comparing three-dimensional sonar and hysteroscopy. Work rationale is that there is a reason to reconsider the status of the diagnostic hysteroscopy to sonohysterography due to evolving technologies, and an improvement in resolution and three dimensional technologies.

DETAILED DESCRIPTION:
Uterine cavity diseases can cause mild to severe symptoms, and may indicate the functional problems of the female reproductive system. Many articles examine the efficacy of diagnostic hysteroscopy compared to sonohysterography in the diagnosis of uterine cavity diseases. Most of the articles are from the last decade, but the subject has been laid aside in the recent years. Antonio Simone Lagana and his group have found that there is 100% correlation in uterine cavity structure between diagnostic hysteroscopy and sonohysterography, and only 78% correlation when it comes to intrauterine fibroids and polyps. Walid El-Sherbiny, MD and his group have found that there is a significant advantage to three-dimensional sonohysterography over two-dimensional in the diagnosis of uterine cavity diseases. No significant difference was observed, and 97% correlation was found, comparing three-dimensional sonar and hysteroscopy. Work rationale is that there is a reason to reconsider the status of the diagnostic hysteroscopy to sonohysterography due to evolving technologies, and an improvement in resolution and three dimensional technologies.

Purpose of the study:

Comparison of the sensitivity, specificity, and the amount of information between diagnostic hysteroscopy and sonohysterography (Two and three-dimensional, in abdominal and vaginal access).

The comparison will be will be made immediately after the completion of diagnostic hysteroscopy test, while using liquid drizzled earlier during the hysteroscopy, in order to simulate sonohysterography which is considered less intrusive and is made As part of standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 70 who were referred by a physician to perform diagnostic hysteroscopy.

Exclusion Criteria:

* refusal to sign a consent form

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
The difference between US and hysteroscopy for the diagnosis and assessment of uterine cavity. | 1 hour
  Comparison of structure of Uterine cavity, Is the uterine cavity normal? Yes/no
The difference between US and hysteroscopy for the diagnosis and assessment of polyps | 1 hour
  Is there a polyp? Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Gad Malinger, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No